CLINICAL TRIAL: NCT06422988
Title: Do Probiotics Reduce The Risk Of Severe Necrotising Enterocolitis (NEC) In Infants Born Before 32 Weeks Gestation? An Observational Study Using Routinely Collected Data.
Brief Title: Do Probiotics Reduce The Risk Of Severe Necrotising Enterocolitis (NEC) In Infants Born Before 32 Weeks Gestation?
Status: Enrolling by invitation | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: University of Nottingham (Other); Newcastle University (Other); Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Cheryl Battersby, Clinical Senior Lecturer, Imperial College London
Other Study IDs: IRAS323099
Record Dates: First submitted 2024-04-24; First posted 2024-05-21 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Enterocolitis, Necrotizing
Keywords: Probiotics
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Probiotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed to probiotics: Receipt of any probiotic in the first 14 days of life. Probiotics to include: Labinic, Proprems probiotic, Acidophillus, Bifidobacterium, Bio-kult, Infloran, LB2.
  To address potential recording error, infants whose NNRD records show minimal (one day) of probiotic exposure will only be classed as exposed if they are cared for in a probiotic unit. Probiotic units are defined as:
  * units who have confirmed that a guideline was in place to provide probiotics to infants born before 32 weeks gestation and that the guideline was in place at any point in the year that the infant was born OR
  * units where more than 50% of the infants eligible to be part of the cohort received probiotics in the six months after the infant was born.
  Interventions: Dietary Supplement: Probiotics
- No probiotic exposure: Did not receive any probiotic in the first 14 days of life.
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Any exposure to probiotics in first 14 days of life
  Other Names: Labinic; Proprems; Acidophillus; Bifidobacterium; Bio-kult; Infloran; LB2

SUMMARY:
Necrotising enterocolitis (NEC) is one of the leading causes of mortality and morbidity in very preterm infants. This study aims to determine whether NEC rates are different between infants who receive probiotics versus infants who do not receive probiotics. The study has a retrospective cohort design and will utilise routinely collected data from the UK National Neonatal Research Database (NNRD). The cohort will comprise all infants born before 32 weeks gestation and cared for in neonatal units in England and Wales between 2016 and 2022. A propensity score matched approach will be used to conduct two comparisons: i) the risk of necrotising enterocolitis (NEC) between who do and those who do not receive probiotics in the first 14 days of life ii) the risk of NEC between babies who receive the two most common probiotic products used in UK units, (Labinic and Proprems).

ELIGIBILITY:
Inclusion Criteria:

* Eligible infants must have been born at less than 32 weeks gestation and be cared for in a English or Welsh unit which contributes data to the National Neonatal Research Database (this includes all NHS neonatal units in England and Wales).
* Infants born in the period January 1st, 2016, to December 31st, 2022 (7 years) will be included.

Exclusion Criteria:

* They have missing data for any of: gestational age at birth, birth weight, year of birth and date of death (for those that died).
* Their NNRD record does not include details of their first admission or begins after Day 3 of life.
* The absolute value of their recorded birthweight for gestational age z score exceeds 4 or is missing.
* They die in the first two postnatal days of life.
* They have a major congenital abnormality

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants born very preterm i.e. before 32 weeks gestation
Sampling Method: Non-Probability Sample
Enrollment: 48000 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Severe necrotising enterocolitis (NEC) | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  NEC confirmed at surgery or postmortem or listed as a cause of death

SECONDARY OUTCOMES:
Necrotising enterocolitis (NNAP definition) | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  NEC diagnosed at postmortem or NEC diagnosed during surgery or NEC diagnosed using clinical and radiographic features (where the infant has at least one clinical feature (bilious gastric aspirate or emesis, abdominal distension, occult, gross blood in stool) and at least one radiographic feature (pneumatosis, hepato-biliary gas, pneumoperitoneum)).
Pragmatically defined NEC | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  Infants who had a recorded diagnosis of necrotising enterocolitis and received at least 5 consecutive days of antibiotics whilst also nil by mouth
Late onset sepsis | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  HQIP NNAP case definition
Pragmatically defined late onset sepsis | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  Growth of any organisms that appear in the NNAP lists of "Clearly pathogenic organisms" and "Other organisms"
Survival to discharge home | On date of discharge from final neonatal unit, assessed up to 24 months
Survival without severe NEC or late onset sepsis (LOS) | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  LOS is defined according to the Healthcare Quality Improvement Partnership (HQIP) National Neonatal Audit Programme (NNAP) case definition i.e. blood stream or cerebrospinal fluid confirmed pure growth in culture after first three days of life
Survival without any NEC | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  NEC is defined as per the NNAP definition
Brain injury | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  Either left or right grade 3 or higher intra-ventricular haemorrhage or cystic periventricular leukomalacia
Treated retinopathy of prematurity | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  Defined as cryotherapy, laser therapy or injection of anti-vascular endothelial growth factor therapy for ROP in either or both eyes
Stage of retinopathy of prematurity | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
Bronchopulmonary dysplasia | 36 weeks postmenstrual age
  Defined as any respiratory or ventilatory support or supplemental oxygen at 36 weeks postmenstrual age
Severe bronchopulmonary dysplasia | 36 weeks postmenstrual age
  Defined as ventilation via endotracheal tube or trachestomy, and excluding non-invasive support or CPAP, at 36 weeks postmenstrual age
Length of stay | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  Number of days between first neonatal unit admission and final neonatal unit discharge for surviving infants
Time to full feeds | Before discharge from final neonatal unit
  Defined as the number of days until an infant is recorded as not requiring any parenteral nutrition or fluid (i.e. no parenteral nutrition or intravenous dextrose)
Growth | 36 weeks corrected gestational age
  Weight for post-menstrual age standard deviation score

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol available now. Analysis code will be available after publication of results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT06422988/Prot_SAP_001.pdf